CLINICAL TRIAL: NCT06016725
Title: E-PROOF: E-Intervention for Protein Intake and Resistance Training to Optimize Function
Brief Title: Online Dietary and Resistance Training to Improve Physical Function in Older Cancer Survivors, E-PROOF Trial
Acronym: E-PROOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jessica Krok-Schoen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-22329; NCI-2023-04622 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21AG078258 (NIH)
Record Dates: First submitted 2023-06-26; First posted 2023-08-30 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage I Prostate Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Prostatic Neoplasms | interventions — Nutrition Assessment; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (nutritional counseling, resistance training) (Experimental): Patients participate in online nutritional counseling over 30 minutes in weeks 1, 3, 5, 7, 9, and 11, and participate in online resistance training sessions weekly over 30 minutes in weeks 1-6 and biweekly at weeks 8, 10, and 12. Patients also receive educational materials at baseline.
  Interventions: Other: Exercise Intervention; Other: Informational Intervention; Other: Nutritional Assessment; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm 2 (educational materials) (Active Comparator): Patients receive educational materials at baseline.
  Interventions: Other: Informational Intervention; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Exercise Intervention — Participate in online resistance training sessions
  Arms: Arm 1 (nutritional counseling, resistance training)
Other: Informational Intervention — Given educational materials
Other: Nutritional Assessment — Participate in online nutritional counseling
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
  Arms: Arm 1 (nutritional counseling, resistance training)
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial tests the feasibility, acceptability, and preliminary effectiveness of online dietary and resistance training to improve physical function in older (greater than or equal to 65-years old) cancer survivors. Declines in adequate protein and calorie intake results in faster loss of muscle mass and physical functioning in older adults. A novel approach to improving physical function in older cancer survivors (OCS) is to utilize online, tailored education and counseling from registered dietitians and exercise scientists, to improve dietary intake (protein intake, diet quality) and participation in resistance exercise. The purpose of this study is to help researchers learn whether an online dietary and resistance training intervention improves diet, exercise, physical function, and health outcomes in OCS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility and acceptability of implementing a 12-week online dietary and resistance training randomized trial with 70 older cancer survivors.

II. Examine the preliminary efficacy of this 12-week online dietary and resistance training intervention with the intervention participants.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients participate in online nutritional counseling over 30 minutes in weeks 1, 3, 5, 7, 9, and 11, and participate in online resistance training sessions weekly over 30 minutes in weeks 1-6 and biweekly at weeks 8, 10, and 12. Patients also receive educational materials at baseline.

ARM 2: Patients receive educational materials at baseline.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* >= 65 years of age
* A primary diagnosis of stage I-III breast, colorectal, and prostate cancer
* Completion of primary curative treatment
* Reported at least 1 physical function limitation on the RAND-36 Physical Function Subscale (PFSS) ("limited a little", "limited a lot")
* No evidence of progressive disease or second cancers
* Community-dwelling
* Able to provide consent

Exclusion Criteria:

* Currently receive cancer treatment (e.g., chemotherapy, radiation)
* Have liver and/or renal disease limiting their protein intake
* Are under the care of a Registered Dietician (RD)/nutritionist
* Participating in other diet/exercise interventions
* Consume protein supplements
* Have contraindications to unsupervised exercise (e.g., walker/wheelchair use)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Krok-Schoen, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 (Nutritional Counseling, Resistance Training) | Arm 2 (Educational Materials)
Started | 38 | 37
Completed | 30 | 33
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Nutritional Counseling, Resistance Training) | Arm 2 (Educational Materials) | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 38 | 37 | 75
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [67 to 72] | 70 [67 to 76] | 70 [67 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 30 | 33 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75
Short Physical Performance Battery [Mean (Full Range); unit: units on a scale] — The physical performance assessment, Short Physical Performance Battery (SPPB), will measure physical function at baseline, end-of-study, and follow-up. The SPPB includes three lower extremity physical performance measures (standing balance, five consecutive chair rises, 4-meter gait walk at usual pace), all summed, to assess lower extremity strength. Summary scores range from 0 to 12, with higher scores denoting higher physical function.
  units on a scale | 9.2 [5 to 12] | 9.1 [6 to 12] | 9.1 [5 to 12]
Grip strength [Mean (Standard Deviation); unit: kg] — Handgrip strength will be measured at baseline, end-of-study, and follow-up in both hands using a hydraulic grip strength dynamometer (Jamar Model 7498). Three trials with brief pauses will be conducted for each hand and the mean score of the six trials will be used as the mean handgrip score (in kgs).
  kg | 27.3 (4.8) | 26.8 (4.3) | 27.0 (4.5)
Diet History Questionnaire III [Mean (Inter-Quartile Range); unit: units on a scale] — Dietary quality was assessed at baseline and end-of-study by the National Cancer Institute's Diet History Questionnaire III (DHQIII).The DHQIII assesses Healthy Eating Index-2015 (HEI-2015) total and individual component scores (e.g., protein) and average daily nutrient intakes, according to the dietary guidelines. Scores can range from 0-100, with higher scores denoting higher dietary quality.
  units on a scale | 66.9 [60.3 to 73.6] | 65.8 [59.2 to 72.5] | 66.3 [59.2 to 73.6]
Godin leisure time exercise [Mean (Standard Deviation); unit: units on a scale] — Self-reported resistance exercise, vigorous, moderate, and mild exercise was assessed using the revised version of The Godin-Shephard Leisure-Time Exercise Questionnaire modified to specifically capture self-reported resistance exercise participation. Scores on the Godin can range from 0-14 units (insufficiently active), 14-23 units (moderately active), or 24 or more units (active). There is no scoring limit.
  units on a scale | 43 (9.8) | 42 (9.2) | 43 (9.6)
RAND-36 [Mean (Standard Deviation); unit: units on a scale] — RAND-36 Health Status Measure is comprised of 8 subscales assessing multiple aspects of HRQoL. Physical and mental component summaries are created. All scores range from 0-100, with 100 as the highest. Changes of ≥5 points on the component scores are considered clinically relevant
  units on a scale | 64.2 (19.2) | 63.0 (21.3) | 63.6 (20.1)
Self-efficacy for diet and exercise [Mean (Standard Deviation); unit: units on a scale] — Baseline and end-of-study self-efficacy for diet and resistance training were measured by: "How sure are you that you could do exercises to make your body stronger for 15 minutes, 3 days a week?" and "How sure are you that you could improve your diet?" A 10-point Likert response scale, ranging from a score of 1 (completely uncertain) to 10 (completely certain), was used.
  units on a scale | 7.6 (2.1) | 8.6 (2.3) | 8.08 (2.2)
Self-regulation for diet and exercise [Mean (Standard Deviation); unit: units on a scale] — Baseline and end-of-study self-regulation for diet and exercise will be measured by the 12-item Dietary Self-Regulation Scale and the 12-item Exercise Self-Regulation Scale. Questions are on a 5-item Likert scale 1-5, never to strongly agree. Each self-regulation scale sums the scores for each item so the scores can range from 12-60, with higher scores denoting higher self-regulation.
  units on a scale | 35.7 (9.8) | 35.6 (10.3) | 35.7 (9.9)
eHealth Literacy Scale [Mean (Standard Deviation); unit: units on a scale] — The 8-item eHealth Literacy Scale (eHEALS) measured knowledge, comfort, and perceived skills of engaging in eHealth at baseline and end-of-study. A 5-point Likert scale (strongly disagree to strongly agree) was used. The total summed scores range from 8-40, with higher scores indicating higher self-perceived ehealth literacy.
  units on a scale | 33.4 (5.4) | 32.3 (6.9) | 32.8 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Physical Function at End-of-intervention
Description: Measured by the Short Physical Performance Battery (SPPB) score. The SPPB score is a continuous variable, collected as the total score ranging from 0-12, higher scores denote higher physical function. Values reported are at the end-of-intervention.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
score on a scale | 9.2 (2.2) | 9.1 (2.3)

2. Secondary Outcome: Satisfaction of the Delivery Method and Information Provided by Nutrition and Exercise Counseling Sessions
Description: Percentage of participant satisfaction ("satisfied" and "very satisfied") measured by a 5-item Likert-scale questionnaire. Scores range from 1-5, with 5 being the highest score of satisfaction.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
score on a scale | 5 [1 to 5] | 5 [1 to 5]

3. Secondary Outcome: Study Accrual Rate
Description: Will be calculated by dividing the number of potential participants that passed screening by the total number of participants started in the study after appropriate informed consent procedures.
Time Frame: assessed during the 12 month recruitment period
Population: The number of participants analyzed represents all potential older cancer survivors (OCS) contacted and assessed for eligibility for participation in the study.
Measure: Number; unit: percentage of participants
Groups:
- All potential participants: Potential participants (older (age ≥65) cancer survivors) were assessed for eligibility in the study.
Arm/Group | All potential participants
Number analyzed (Participants) | 324
percentage of participants | 23.1

4. Secondary Outcome: Study Retention Rate
Description: calculated by dividing the total number of participants initiated by total number of participants in the study. Retention goal for this trial is 80%. If 80% (56/70) of participants are retained at end-of-study, the retention goal for this trial will be achieved. Overall retention rates and associated 95% confidence intervals will be reported.
Time Frame: End-of-study, up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
Participants | 30 | 33

5. Secondary Outcome: Study Adherence Rate
Description: Participants were determined to be adherent if they attend >= 80% of the online intervention sessions. Overall adherence rates and associated 95% confidence intervals were reported.
Time Frame: end-of-intervention, at 12 weeks
Population: Percentage of Participants who Attended >= 80% of the Intervention Sessions
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
percentage of participants | 97 | 95

6. Secondary Outcome: Grip Strength
Description: Handgrip strength (absolute value at the end of the intervention) was measured in both hands using a hydraulic grip strength dynamometer. This is measured in kgs.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Standard Deviation); unit: kgs
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
kgs | 28.6 (5.2) | 28.3 (4.8)

7. Secondary Outcome: Dietary Quality
Description: Dietary quality was assessed by the National Cancer Institute's Diet History Questionnaire III using the Healthy Eating Index score ranging 0-100, with higher scores meaning higher diet quality. Absolute value at end-of-intervention was assessed using the Healthy Eating Index score.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
score on a scale | 69.3 [63 to 76] | 68.1 [61 to 75]

8. Secondary Outcome: Percentage of Participants Who Completed Resistance Exercises
Description: Self-reported resistance exercise (% yes) was assessed using the revised version of The Godin-Shephard Leisure-Time Exercise Questionnaire modified to specifically capture self-reported resistance exercise participation. If a participant denoted "yes" to the question: did During a typical 7-Day period (a week), did you participate in resistance exercise for more than 15 minutes during your free time? Percentages denote the percentage of the study subjects who participated in resistance training at end of intervention.
Time Frame: end-of-intervention, at 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
percentage of participants | 97 | 65

9. Secondary Outcome: Health-related Quality of Life (HRQoL)
Description: RAND-36 Health Status Measure is comprised of 36 items which automatically create 8 subscales assessing multiple aspects of HRQoL. All scores range from 0-100, with 100 as the highest HRQoL. The main HRQoL subscale reported is the general health HRQoL subscale. Mean scores of general HRQoL for end-of-intervention are reported.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
score on a scale | 53.8 (18.9) | 60.1 (19.1)

10. Secondary Outcome: Self-efficacy
Description: Self-efficacy was measured at the end of intervention via a 0-10 confidence scale rating the confidence of making exercise and diet changes in one's life, with 0 meaning not confident, 10 meaning very confident.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
score on a scale | 9.47 (2.1) | 8.97 (1.9)

11. Secondary Outcome: Technology Competency
Description: The 8-item eHealth Literacy Scale measured knowledge, comfort, and perceived skills of engaging in eHealth at end-of-intervention. A 5-point Likert scale was used, with possible scores ranging from 8 to 40. Higher scores indicate higher ehealth literacy.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
score on a scale | 33.9 [27 to 40] | 33.2 [26 to 40]

12. Secondary Outcome: Anthropometry Body Weight in Kilograms
Description: At end-of-intervention, participant's body weight was assessed in kilograms.
Time Frame: end-of-intervention, at 12 weeks
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
kg | 28 [26 to 32] | 29 [24 to 33]

13. Secondary Outcome: Anthropometry Height in Inches
Description: At end-of-intervention, participants' height was assessed using height in centimeters.
Time Frame: end-of-intervention, at 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
cm | 165.2 (5.2) | 166.1 (4.8)

14. Secondary Outcome: Anthropometry Measuring Waist Circumference in Centimeters
Description: At end-of-intervention, participants' waist circumference was assessed in centimeters.
Time Frame: end-of-intervention, at 12 weeks
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Arm 1 (nutritional counseling, resistance training) | Arm 2 (educational materials)
Number analyzed (Participants) | 38 | 37
cm | 100 [90 to 110] | 101 [89 to 113]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each of the participant's in-person data collection events (baseline, 12 weeks, and 24 weeks). Also participants could contact the study team at any time.
Description: Not different than the definition from clinicaltrials.gov definitions.
Arm/Group | Arm 1 (Nutritional Counseling, Resistance Training) | Arm 2 (Educational Materials)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT06016725/Prot_SAP_000.pdf